CLINICAL TRIAL: NCT03524859
Title: Comparative Analysis of Outcome Measures From Sit-to-stand Test Between Cystic Fibrosis and Healthy Subjects.
Brief Title: Evaluation of Sit-to-stand Test in Patients With Cystic Fibrosis and Matched Controls.
Acronym: STS-CF
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Diego Ruiz-Cárdenas, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: UCMurcia
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Sit-to-stand; Lung Function; Handgrip; Walking Speed; Power; Velocity; Gait Speed; Chair rise
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: Cystic fibrosis participants without experience on endurance or resistance training will be analyzed through a test battery and lung function test.
- Healthy Subjects: Healthy matched control group without experience on endurance or resistance training will be analyzed through a test battery.

SUMMARY:
Introduction: In recent years, since the discovery of the cystic fibrosis (CF) transmembrane conductance regulator gene in human skeletal muscle, there appears to be growing interest in the measurement of muscle function in CF. One of the most used test in other chronic pulmonary diseases is the Sit-to-Stand test (STS) which consists of simply getting up from a chair. Although the main result of the STS test is the time developed during the task, the velocity and power generated during the task are considered very important variables to detect the functional decline. However, from our knowledge, no study has previously analyzed the differences in time, velocity and muscle power developed during the STS test in patients with CF and their respective healthy controls.

Objectives: To compare the values gained from handgrip strength, walking speed and STS test (time, velocity, and muscle power) in a group of patients with CF and their respective healthy controls, and to analyze if these differences (if any) are associated with lung function in patients with CF.

Methods: Cross-sectional study with a sample of 60 participants (30 patients diagnosed with CF and 30 healthy subjects) between 18-65 years old. The STS test will be measured through slow-motion video recording with a smartphone device (240 images per second) which will report the time, velocity and power generated during the test. Walking speed and handgrip strength will be also measured. Additionally, the relationship between the variables obtained during the test and the lung function of patients with CF will be analized.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis clinically stable; without experience on endurance or resistance training; no receiving long-term oxygen therapy.
* Healthy matched controls; without experience on endurance or resistance training.

Exclusion Criteria:

* Using psychotropic medications; concomitant neurological, cardiovascular, metabolic, rheumatic or vestibular diseases; physical disabilities that impaired locomotion or chair rise; orthopedic problems; or a history of musculoskeletal system operations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cystic fibrosis will be recruited from the Cystic Fibrosis Association of Murcia, Spain. Additionally, a non-probabilistic sample from healthy subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Sit-to-stand time | Cross-sectional baseline (non intervention)
  The time to complete the sit-to-stand test will be measured using a smartphone (Sit-to-stand App version 1.1) installed on an iPhone 6 running iOS 11 (Apple Inc., USA).
  To execute the test, subjects will sit on a rigid chair with their arms crossed over their chest with the hip, knee and ankle joints at approximately 90 degrees. The subjects will be instructed to stand-up as fast as possible. Participants will complete three STS repetitions to complete the test while standing without footwear.
Sit-to-stand velocity | Cross-sectional baseline (non intervention)
  The vertical velocity generated by the participants during the sit-to-stand test will be measured using a smartphone (Sit-to-stand App version 1.1) installed on an iPhone 6 running iOS 11 (Apple Inc., USA).
  To execute the test, subjects will sit on a rigid chair with their arms crossed over their chest with the hip, knee and ankle joints at approximately 90 degrees. The subjects will be instructed to stand-up as fast as possible. Participants will complete three STS repetitions to complete the test while standing without footwear.
Sit-to-stand power | Cross-sectional baseline (non intervention)
  The leg power generated by the participants during the sit-to-stand test will be measured using a smartphone (Sit-to-stand App version 1.1) installed on an iPhone 6 running iOS 11 (Apple Inc., USA).
  To execute the test, subjects will sit on a rigid chair with their arms crossed over their chest with the hip, knee and ankle joints at approximately 90 degrees. The subjects will be instructed to stand-up as fast as possible. Participants will complete three STS repetitions to complete the test while standing without footwear.

SECONDARY OUTCOMES:
Handgrip strength | Cross-sectional baseline (non intervention)
  Handgrip testing will be performed in standing position with the arm at the side and the forearm and wrist placed into neutral. Using a digital hand dynamometer, subjects will squeez the device maximally. The test will be repeated two times on both the right and left hand with 30-s of rest between trials of the same hand. The greater of the two trials from the right and left side will be used and added together to give overall handgrip strength.
Walking speed | Cross-sectional baseline (non intervention)
  Self-selected walking speed will be determined by having participants walk at a pace they consider 'normal walking speed' over a distance of 8 m on a non-carpeted floor. To account for the time it will take participants to accelerate and decelerate, markers will be provided 2 m before and after the measured distance. Therefore, the total timed distance will be 4 m. The timed walking test will be completed twice to promote familiarity and improve accuracy.
Lung function | Cross-sectional baseline (non intervention)
  Lung function will be measured with a calibrated spirometer by a experimented nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Diego Ruiz-Cárdenas, PT, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Cystic Fibrosis Association, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruiz-Cardenas JD, Rodriguez-Juan JJ, Smart RR, Jakobi JM, Jones GR. Validity and reliability of an iPhone App to assess time, velocity and leg power during a sit-to-stand functional performance test. Gait Posture. 2018 Jan;59:261-266. doi: 10.1016/j.gaitpost.2017.10.029. Epub 2017 Oct 31. PMID 29102856